CLINICAL TRIAL: NCT00175747
Title: A Randomized Phase IIb Trial of Pulmicort Turbuhaler (Budesonide) in People With Dysplasia of the Bronchial Epithelium
Brief Title: A Phase IIb Trial of Pulmicort Turbuhaler (Budesonide)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USPHS Grant N01-CN85188
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Lung Cancer
Keywords: dysplasia; lung cancer; chemoprevention
MeSH Terms: conditions — Lung Neoplasms

INTERVENTIONS:
Drug: Inhaled Budesonide 800 µg twice daily

SUMMARY:
Studies in animals suggest that inhaled budesonide may prevent the occurrence of lung cancer. We conducted a clinical trial to determine the effects of inhaled budesonide in smokers who had precancerous lesions in the breathing tubes (i.e. bronchial dysplasia.

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer death worldwide: the mortality rate of lung cancer exceeds that of colon, breast, and prostate cancers combined. Former heavy smokers retain an elevated risk for lung cancer even years after they stop smoking. Given the large number of current and former smokers and the increasing incidence of lung cancers among women, lung cancer will remain a major health issue for the next several decades.

One potential strategy to inhibit the development of invasive cancer in those who are at risk of developing lung cancer is to use chemopreventive agents that can regress existing intraepithelial neoplastic lesions, prevent the progression of these lesions to cancer, or prevent the development of new lesions.

We performed a randomized, double-blind, placebo-controlled, phase IIb clinical trial to determine the efficacy and safety of inhaled budesonide (Pulmicort Turbuhaler) as a chemopreventive agent in smokers with premalignant lesions in their bronchial epithelia. The primary end point was change in the histopathologic grade on repeat biopsy of the same sites at the end of 6 months. The secondary end points of this study aimed to gather additional insight into the potential effects of budesonide on the central bronchial epithelial lung compartment, on the peripheral lung that could not be directly assessed through bronchoscopic biopsy, and on drug effect biomarkers that reflect the ability of inhaled budesonide to reach its target. Thus, the balance between proliferation and apoptosis was examined through immunohistochemical analysis of the expression of the proliferative marker MIB-1 and the antiapoptotic protein BclII. Expression of the tumor suppressor p53, which functions to maintain the integrity of the human genome, is a major determinant of cell survival, is frequently mutated in lung cancer, and was assessed in bronchial biopsies. Examination of peripheral pulmonary nodules via spiral computed tomography (CT) was performed to assess, for the first time, the potential usefulness of spiral CT in response to chemopreventive interventions. Finally, prostaglandin E2 (PGE2), a prostaglandin derived from arachidonic acid metabolism whose synthesis is inhibited by glucocorticoids, was measured in the bronchoalveolar lavage fluid.

Study subjects were recruited using television programs, radio broadcasts, and local newspapers between June 1, 2000, and November 1, 2001. Eligibility included age > 40 years, smoking history of 30 pack-years, and normal organ function. Sputum samples were obtained using simultaneous high-frequency chest wall oscillation with a ThAIRapy Vest (Advanced Respiratory, Inc., St. Paul, MN) and inhalation of 3% hypertonic saline from an ultrasonic nebulizer for 12 minutes. The subjects were instructed to cough intermittently during the induction procedure and for at least 2 hours afterward to produce sputum samples. The sputum samples were fixed in 50% etomidate, cytospun onto glass slides, and stained with Feulgen-thionin. The DNA content, the size, shape, and DNA distribution of at least 3000 epithelial cell nuclei per sample were measured using automated high-resolution image cytometry (Cyto-Savant system; Perceptronix Medical, Inc., Vancouver, British Columbia, Canada; refs. 13 , 14 ). Cells were classified as either epithelial, inflammatory, or pyknotic based on these features, and an experienced cytotechnologist confirmed the automated classifications. Diploid DNA had a DNA index of 1.0. Atypia was defined as the presence of more than or equal to five cells having a DNA index > 1.2. This criterion was based on a retrospective analysis of 1885 apparently healthy volunteer smokers who underwent sputum quantitative cytometry as part of the Lung Health Study at the British Columbia Cancer Agency since 1990. Participants were followed by repeat chest X-ray and autofluorescence bronchoscopy if they were in a National Cancer Institute-sponsored chemoprevention trial or through the British Columbia Cancer Registry and the Medical Services Plan Hospital Registry. Using the threshold of more than or equal to five cells with a DNA index > 1.2, the sensitivity of detecting lung cancer in the initial screening or on follow-up was 94%, with a specificity of 38% after a mean follow-up of 3.2 years. This threshold was adopted in the current study to identify smokers with the highest risk for lung cancer for bronchoscopy.

Autofluorescence bronchoscopy was performed in subjects with sputum atypia who agreed to undergo bronchoscopy to localize areas of dysplasia using the LIFE-Lung device (Xillix Technologies Corp., Richmond, British Columbia, Canada). Biopsy samples were taken from areas with abnormal fluorescence that were at least 1.2 mm in size, as well as from at least two control areas of normal fluorescence. The median number of biopsy samples obtained per subject was 6 (range, 4-14 samples). Bronchoalveolar lavage was performed using standard techniques. The collected fluid (30 mL per participant) was immediately placed at 4°C, and a differential cell count was obtained within 1 hour of collection. The fluid was separated from the cells by centrifugation and frozen at -160°C for subsequent PGE2 assays.

The biopsy samples were fixed in buffered formalin, embedded in paraffin, and serially sectioned. H&E-stained sections were systematically reviewed by two pathologists who were blinded to intervention assignments (J. leRiche, A. Gazdar). All biopsy samples were classified into one of the following seven groups (normal, basal cell hyperplasia, metaplasia, mild/moderate/severe dysplasia, or carcinoma in situ) according to WHO criteria. Because individual biopsies frequently contained more than one histologic cell type, the diagnosis was based on the most advanced histology present.

The two pathologists resolved minor (i.e., one grade) differences in sample classification by telephone consultation. If the histopathology diagnosis differed by two or more grades, both pathologists reviewed the slides again and, if necessary, reached a consensus diagnosis after verbal communication by phone or e-mail.

One hundred fifty-one subjects (27% of subjects who underwent bronchoscopy) had one or more sites of bronchial dysplasia with a surface diameter > 1.2 mm (i.e., greater than the size of a bronchial biopsy using standard biopsy forceps). Only subjects with dysplastic lesions > 1.2 mm were enrolled onto the chemoprevention trial to minimize the effect of mechanical removal of these lesions by the biopsy procedure.

Participants were randomly assigned to receive either budesonide (Pulmicort Turbuhaler; AstraZeneca, Lund, Sweden) at a dose of 800 µg twice daily by inhalation or placebo for 6 months. The placebo turbuhalers were identical to the ones containing the active drug. Randomization was stratified according to smoking status (current versus former) and gender. All study personnel were blinded to the study codes, as was confirmed by independent review.

The participants were interviewed monthly for compliance and drug-related adverse events. Compliance was determined from a drug diary and from estimation of the number of doses remaining in the turbuhaler. Toxicity was monitored according to the National Cancer Institute Common Toxicity Criteria, version 2.0.10 Dose modification was performed for any grade 2 toxicity or for evidence of cortisol suppression (ante meridiem (AM) plasma cortisol < 140 nmol/L/L). For grade 3 or 4 toxicity, therapy was discontinued until toxicity resolved to grade 1 or less. At that time, the use of the study drug was resumed with a 75% dose reduction.

All participants underwent a second fluorescence bronchoscopy with bronchoalveolar lavage after 6 months on study medication and biopsies were obtained from the same sites biopsied at baseline. Biopsy samples were also taken from new areas that displayed abnormal fluorescence. The bronchoscopist was blinded to the intervention assignment.

Current smokers were encouraged to stop smoking and were invited to take part in the Fresh Start Program at the British Columbia Cancer Agency. The Clinical Investigations Committees of the British Columbia Cancer Agency and the University of British Columbia approved this study. Written informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* age > 40 years; smoking history of 30 pack-years or more; normal organ function; sputum atypia

Exclusion Criteria:

* general debility that would prevent completion of 6 month follow-up; existing cancer diagnosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2000-01; Study Completion 2002-12

PRIMARY OUTCOMES:
Rate of progression of bronchial dysplasia

SECONDARY OUTCOMES:
Number of pulmonary nodules on thoracic CT scanning and BCL-2 and p53 expression in the bronchial epithelial cells.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, MD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Lam S, leRiche JC, McWilliams A, Macaulay C, Dyachkova Y, Szabo E, Mayo J, Schellenberg R, Coldman A, Hawk E, Gazdar A. A randomized phase IIb trial of pulmicort turbuhaler (budesonide) in people with dysplasia of the bronchial epithelium. Clin Cancer Res. 2004 Oct 1;10(19):6502-11. doi: 10.1158/1078-0432.CCR-04-0686. PMID 15475437